CLINICAL TRIAL: NCT00564811
Title: Effect of Agaricus Blazei (Murrill) ss. Heinemann (Sun Mushroom) on the Nutritional State and Liver Biochemistry in Hepatitis C Patients.
Brief Title: Effect of Agaricus Blazei (Murrill) ss. Heinemann (Sun Mushroom)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-03
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis C; Nutritional Status; Hepatitis, Viral, Human
Keywords: Agaricus blazei (Murrill) ss. Heinemann,; Hepatitis C; Nutritional status; Liver Function Tests; Antiviral Agents
MeSH Terms: conditions — Hepatitis C; Hepatitis, Viral, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G1 (No Intervention)
- G2 (Experimental)
  Interventions: Dietary Supplement: Agaricus blazei (Murrill) ss. Heinemann (sun mushroom)

INTERVENTIONS:
Dietary Supplement: Agaricus blazei (Murrill) ss. Heinemann (sun mushroom) — Agaricus blazei powder, 10 grams/day, for 5 months
  Arms: G2

SUMMARY:
The aim of the study was to verify the influence of Agaricus blazei (Murrill) ss. Heinemann (A. blazei) on the evolution of nutritional state and liver function in hepatitis C patients.

DETAILED DESCRIPTION:
Ten patients were studied (5 - GI - not taking A. blazei - and 5 - G2 - taking A. blazei), from both sexes, with positive Anti-VHC and a healthy nutritional state, admitted into in the viral hepatitis ward. Diagnosis and treatment for hepatitis C concurred with the regulations of the Ministry of Health and nutritional evaluation was performed in 3 moments according to anthropometrical, bioimpedance, biochemical and dietary standards, with duration of 6 months. The consumption of A. blazei (10g/day) in dehydrated powder was concomitant with antiviral therapy (conventional or pegylated interferon associated with ribavirin) with duration of 5 months.

ELIGIBILITY:
Inclusion Criteria:

* To have been informed and signed adequately the free and clarified assent
* Initiating the anti-viral treatment (interferon or pegylated interferon associate the ribavirin)
* Age: 24-70 years
* Gender :both the gender
* Race : all races
* To present serology positive to the anti-VHC ELISA
* To present genotype type 1,2,or 3
* Body mass index- >18,5 e < 35kg /m2
* Conditions full to the ORAL ingestion

Exclusion Criteria:

* Don't agree to the project or don't have signed the term of clarified free assent
* Restriction for oral ingestion
* The existence of surface of antigen of the hepatitis B virus(Ag HBs)
* The existence of antibody for the human immunodeficiency virus
* To be enclosed in another project of research or form of treatment
* Pregnant women
* Suckles
* Cirrhosis
* Patients with hepatitis auto-imune.

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-03; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Measure: influence of Agaricus blazei (Murrill) ss. Heinemann on the evolution of nutritional state and liver function in hepatitis C patients. Time Frame: six months | Time Frame: six months

CONTACTS AND LOCATIONS:
Overall Officials: Caramori A Carlos, MD, PhD, Study Chair — Botucatu Medicine School - Sao Paulo State University
Locations (1):
- Internal Medicine Department, Botucatu School of Medicine, São Paulo State University - UNESP, Botucatu, São Paulo, Brazil